CLINICAL TRIAL: NCT05398835
Title: An Online Intervention Promoting Home-based HIV Self-testing Among Men Who Have Sex With Men in Hong Kong During the COVID-19 Pandemic
Brief Title: Promoting HIV Self-testing Among MSM During COVID-19 Pandemic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Zixin Wang, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: KPF19HLF16
Record Dates: First submitted 2022-05-30; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Health Behavior
Keywords: HIV testing; HIV self-testing
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Online interventions promoting home-based HIV self-testing
  Interventions: Behavioral: Online interventions promoting HIV self-testing

INTERVENTIONS:
Behavioral: Online interventions promoting HIV self-testing — 1) viewing an online video promoting HIVST, 2) visiting the project webpage containing demonstration video of how to use HIVST kits, information about local HIV epidemic and benefits of HIV testing and HIVST, and a discussion forum containing positive feedback of HIVST users, and 3) having access to a chargeable HIVST services implemented by the CBO

SUMMARY:
A community-based organization (CBO) recruited Chinese-speaking men who have sex with men who are HIV-negative or unknown sero-status through multiple channels in Hong Kong, China.

Participants first complete a baseline telephone survey, and then receive the following health promotion components: 1) viewing an online video promoting HIVST, 2) visiting the project webpage containing demonstration video of how to use HIVST kits, information about local HIV epidemic and benefits of HIV testing and HIVST, and a discussion forum containing positive feedback of HIVST users, and 3) having access to a chargeable HIVST services implemented by the CBO.

All participants are invited to complete a follow-up telephone survey six months after completion of the baseline survey.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above
* Having access to internet
* Anal intercourse with at least one man in the past six months
* Willing to complete telephone follow-up survey at Month 6

Exclusion Criteria:

* Self-reported to be HIV positive

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
HIV testing | 6 months
  Uptake of any type of HIV testing
HIV self-testing | 6 months
  Uptake of any type of home-based HIV self-testing

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Health Behaviours Research, the Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No